CLINICAL TRIAL: NCT00824122
Title: Genetic Polymorphisms Associated With Histamine Disposition in Children With Vancomycin Associated Red Man Syndrome (RMS)
Brief Title: Vancomycin Associated Red Man Syndrome (RMS)
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Katherine Berry Richardson Foundation (Unknown)
Responsible Party: Principal Investigator, Angela Myers, Assistant Professor of Pediatrics, Children's Mercy Hospital Kansas City
Other Study IDs: 10914
Record Dates: First submitted 2009-01-14; First posted 2009-01-16 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Red Man Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Frozen blood has been maintained for future genetic studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Children greater than 6 months receiving at least one dose of Vancomycin and Red Man Syndrome
- 2: Children greater than 6 months receiving at least one dose of Vancomycin and has not had Red Man Syndrome

SUMMARY:
This study proposes to identify patients who developed RMS with vancomycin infusion, and determine presence or absence of variant alleles involved in histamine biotransformation. The implications of this study are important, as identification of variant alleles in these patients, may alter the current standard of care for vancomycin infusions.

The hypothesis of this study is that the development of red man syndrome (RMS) during receipt of intravenous vancomycin is associated with the presence of variant alleles for genes involved in the histamine pathway. The primary outcome that will be measured will be the history of RMS and the presence or absence of variant alleles for the genes responsible for histamine metabolism (i.e. histamine n-methyltransferase and diamine oxidase). As a secondary endpoint, the study will also attempt to determine the incidence of RMS in pediatric patients.

DETAILED DESCRIPTION:
Vancomycin has been utilized as an antimicrobial therapeutic agent for serious gram positive infections for more than half a century.The pharmacokinetics of vancomycin has been well studied, and in general there are few side effects from this medication. The most common side effect that occurs with receipt of vancomycin is red man syndrome (RMS), which is also known as red neck, or red person syndrome.1 RMS encompasses a spectrum that ranges from a mild reaction such as flushing, urticarial rash, pruritis, to a severe reaction that includes generalized erythema,intense pruritis, and even hypotension. RMS has been estimated to occur in 5- 50% of hospitalized patients who receive this drug.

RMS is considered an anaphylactoid type of reaction that is due to mast cell degranulation with a concomitant rise in blood histamine levels. The resultant symptomatology varies from mild itching and erythematous rash to a more generalized reaction with hypotension. This reaction has been shown to be modified by pre-treatment with various types of antihistamines including diphenhydramine and cimetidine.

There is now evidence to suggest that altered histamine metabolism contributes to the pathogenesis of various disorders. Histamine is almost exclusively metabolized by the enzymes histamine N-methyltranserase (HNMT)and diamine oxidase (DAO) both of which are polymorphically expressed in people with varying frequencies.HNMT catalyzes the N- methylation of histamine. This is the predominant pathway for histamine metabolism,accounting for 50-80% of its biotransformation. Diamine oxidase (DAO) likely contributes in a significant manner of the remaining metabolism of histamine as only 2-3% of this autocoid is excreted unchanged in the urine. It is plausible that allelic variants of HNMT and/or DAO may contribute to histmaminergic reactions in a given patient with resultant propagation of its pharmacologic effects, and that polymorphically expressed enzymes primarily responsible for terminating the pharmacologic activity of histamine (via biotransformation)may play a crucial role in determining disease phenotype for disorders (e.g., RMS) where histamine is a key mediator.

This is a prospective study that will be conducted over a one year period of time. Eligible patients will be identified by a search of patients who are receiving vancomycin therapy throughout the study period. Chart review/patient interview will then be performed to identify patients who developed symptomatology consistent with RMS while receiving vancomycin infusion. For the purposes of this study, red man syndrome (RMS) will be defined as: erythematous rash, flushing of the face, neck, or torso, itching, or a lowering of systolic or diastolic blood pressure by >10mm/hg. A subset of patients who remained asymptomatic throughout their vancomycin therapy will also be evaluated as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received vancomycin

Exclusion Criteria:

* Patients who have received antihistamines at the time of vancomycin administration or
* Patients who have been on steroids or tricyclic antidepressants within 30 days prior to the vancomycin administration
* People receiving ECMO or have multiorgan failure
* Currently receiving dialysis

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Eligible patients will be identified by a search of patients who are receiving vancomycin therapy throughout the study period. Chart review/patient interview will then be performed to identify patients who developed symptomatology consistent with RMS while receiving vancomycin infusion. For the purposes of this study, red man syndrome (RMS) will be defined as: erythematous rash, flushing of the face, neck, or torso, itching, or a lowering of systolic or diastolic blood pressure by >10mm/hg. A subset of patients who remained asymptomatic throughout their vancomycin therapy will also be evaluated as a control group.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Presence or abscence of genetic polymorphisms in the histamine pathway in patients with vancomycin related RMS. | During Hospital Admission

CONTACTS AND LOCATIONS:
Overall Officials: Angela Myers, MD, MPH, Principal Investigator — Children's Mercy Hosptials and Clinics
Locations (1):
- Children's Mercy Hospital & Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Myers AL, Gaedigk A, Dai H, James LP, Jones BL, Neville KA. Defining risk factors for red man syndrome in children and adults. Pediatr Infect Dis J. 2012 May;31(5):464-8. doi: 10.1097/INF.0b013e31824e10d7. PMID 22327873